CLINICAL TRIAL: NCT07091136
Title: Exploration of Manidipine to Reverse Aortic Valve Calcification by Activating Valvular Osteoclasts in Patients With Severe Calcific Aortic Valvular Disease
Brief Title: Exploration of Manidipine to Reverse Aortic Valve Calcification
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Wuhan Union Hospital
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Calcific Aortic Valve Disease
Keywords: manidipine; Calcific Aortic Valve disease
MeSH Terms: interventions — manidipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- manidipine 10 mg (Experimental): Participants are giving manidipine 10 mg once daily for 12 months, followed by a 3-month safety observation.
  Interventions: Drug: manidipine
- placebo (Placebo Comparator): Participants are giving placebo once daily for 12 months, followed by a 3-month safety observation.
  Interventions: Drug: Placebo
- manidipine 20 mg (Experimental): Participants are giving manidipine 20 mg once daily for 12 months, followed by a 3-month safety observation.
  Interventions: Drug: manidipine

INTERVENTIONS:
Drug: manidipine — study will enrol 100 adults aged 60 to 85 years with MDCT-confirmed mild-to-moderate aortic valve calcification (Agatston score 300-2 000 AU) and preserved left-ventricular ejection fraction to receive manidipine 10 mg, manidipine 20 mg, or matched placebo once daily for 12 months, followed by a 3-month safety observation, with the primary endpoint being the absolute and relative change in aortic valve calcium score at 12 months; secondary endpoints include echocardiographic valve area and transvalvular gradients, six-minute walk distance, peak oxygen uptake, and comprehensive safety outcomes
  Arms: manidipine 10 mg; manidipine 20 mg
Drug: Placebo — study will enrol 100 adults aged 60 to 85 years with MDCT-confirmed mild-to-moderate aortic valve calcification (Agatston score 300-2 000 AU) and preserved left-ventricular ejection fraction to receive manidipine 10 mg, manidipine 20 mg, or matched placebo once daily for 12 months, followed by a 3-month safety observation, with the primary endpoint being the absolute and relative change in aortic valve calcium score at 12 months; secondary endpoints include echocardiographic valve area and transvalvular gradients, six-minute walk distance, peak oxygen uptake, and comprehensive safety outcomes
  Arms: placebo

SUMMARY:
This is a prospective, randomized, comparative, clinical trial conducted by Wuhan Union Hospital that aims to evaluate the efficacy and safety of manidipine compared to placebo in patients with calcific aortic valve disease with mild aortic valve stenosis.

DETAILED DESCRIPTION:
This multicentre, randomized, double-blind, placebo-controlled phase IIb study will enrol 100 adults aged 60 to 85 years with MDCT-confirmed mild-to-moderate aortic valve calcification (Agatston score 300-2 000 AU) and preserved left-ventricular ejection fraction to receive manidipine 10 mg, manidipine 20 mg, or matched placebo once daily for 12 months, followed by a 3-month safety observation, with the primary endpoint being the absolute and relative change in aortic valve calcium score at 12 months; secondary endpoints include echocardiographic valve area and transvalvular gradients, six-minute walk distance, peak oxygen uptake, and comprehensive safety outcomes; the trial is grounded in extensive mechanistic work showing that calcific heart valve disease affects more than 209 million people worldwide-over 25 million in China alone-and that osteoclast deficiency or dysfunction within valvular tissue is a pivotal driver of progressive calcium deposition, with persistent up-regulation of the NLRP3 inflammasome suppressing osteoclastogenesis and the key resorptive enzyme Cathepsin K; through high-content screening of 198 candidate NLRP3 inhibitors and confirmatory concentration-response assays, the investigators identified the fourth-generation dihydropyridine calcium-channel blocker manidipine as uniquely capable of simultaneously down-regulating NLRP3 and up-regulating Cathepsin K, thereby restoring osteoclastic capacity to dissolve pathological calcium deposits and dramatically reducing valvular calcification in murine models; extrapolating these findings to humans, the study seeks to establish manidipine as the first mechanism-based, orally available, cost-effective pharmacotherapy capable of halting or reversing calcific progression, potentially obviating or delaying the need for valve replacement surgery, mitigating the limitations of current mechanical and bioprosthetic options (lifelong anticoagulation, re-calcification, repeat procedures), and ultimately reducing morbidity, mortality, and healthcare expenditure associated with CHVD; rigorous imaging core-lab analysis, blinded adjudication of endpoints by an independent committee, and periodic oversight by a data-safety monitoring board will ensure robustness of findings, while predefined statistical plans employing ANCOVA for the primary endpoint (with baseline calcium score and centre as covariates), mixed-effects models for repeated-measures secondary variables, and survival analysis for clinical events will provide comprehensive efficacy and safety profiles; if the trial demonstrates a clinically meaningful slowing or reversal of calcification alongside an acceptable safety profile, manidipine could rapidly progress to phase III evaluation and, given its established antihypertensive indications and favourable pharmacokinetics, could be repurposed swiftly to address the global unmet need for a pharmacological solution to calcific heart valve disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult ≥ 60 years of age at the time of rescruiting.
* Subject has calcific aortic valve disease with mild to moderate aortic valve stenosis as defined by Doppler echocardiography results: Aortic Valve mean pressure gradient between 10-30 mmHg and Aortic Valve Area ≥ 1.2 and ≤ 2.0 cm2 on TTE within 2 weeks prior to randomization and Cardiac Compute Tomography (CT) test results: aortic valve calcium score (Agatston score) ≥ 200 AU at baseline cardiac CT within 1 month prior to randomization
* Subject provides written informed consent prior to initiation of any study procedures.
* Subject understands and agrees to comply with planned study procedures.

Exclusion Criteria:

* Subject has concomitant moderate or severe mitral or tricuspid valve disease.
* Subject has left ventricular ejection fraction < 50%.
* Subject previous history of aortic valve surgery, pancreatitis, malignant tumor, drug or alcohol abuse.
* Subjects whose alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 2.5 times the upper limit of normal range.
* Subjects who cannot undergo Cardiac CT.
* Pregnant or lactating women.
* Consideration by the investigator, for safety reasons, that the subject is an unsuitable candidate to receive study treatment.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
aortic valve calcification | 3 month later than stop drug giving
  Measure aortic valve calcification Agatston score of participants with CTA.

SECONDARY OUTCOMES:
overall survival | 1 year
  follow up the survival condition after giving drugs
Change in aortic valve stenosis severity | 1 year
  Change in aortic valve stenosis severity as measured by peak transaortic velocity using echocardiography at week 104 as compared to baseline
Time-to-major adverse cardiovascular events | 1 year
  Time-to-major adverse cardiovascular events of cardiac death, non- fatal myocardial infarction, heart failure hospitalization and stroke

IPD SHARING:
Plan to Share IPD: Undecided